CLINICAL TRIAL: NCT01667146
Title: A Multi-centre Randomised Controlled Trial of an Open Lung Strategy Including Permissive Hypercapnia, Alveolar Recruitment and Low Airway Pressure in Patients With Acute Respiratory Distress Syndrome.
Brief Title: Open Lung Ventilation in ARDS: The PHARLAP Trial
Acronym: PHARLAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Halted by the Management Committee after the publication of the ART Trial
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: University College Dublin (Other)
Responsible Party: Principal Investigator, Carol Hodgson, Dr Carol Hodgson, Australian and New Zealand Intensive Care Research Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANZIC-RC/AD002 Version 8
Record Dates: First submitted 2012-08-12; First posted 2012-08-17 (Estimated); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-02

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PHARLAP ventilation group (Experimental): PHARLAP mechanical ventilation strategy
  Interventions: Other: PHARLAP mechanical ventilation strategy
- Control group ventilation (Active Comparator): Control group mechanical ventilation strategy
  Interventions: Other: Control group mechanical ventilation strategy

INTERVENTIONS:
Other: PHARLAP mechanical ventilation strategy — Pressure control ventilation to maintain tidal volume 4-6 ml/kg and plateau pressure ≤ 30 cmH2O while tolerating respiratory acidosis if pH > 7.15; daily staircase recruitment manoeuvre and individualised PEEP titration.
  Arms: PHARLAP ventilation group
Other: Control group mechanical ventilation strategy — Mechanical ventilation based on the ARDSnet protocol using volume control ventilation with tidal volume 6 ml/kg, plateau pressure ≤ 30 cmH2O and FiO2/PEEP titration according to a FiO2/PEEP/oxygen saturation combination chart. This has been modified for Australian and New Zealand practice to allow pressure control and pressure support ventilation.
  Arms: Control group ventilation

SUMMARY:
Some people develop the condition called acute respiratory distress syndrome (ARDS). This is a condition where the lungs have become injured from one of a number of various causes, and do not work as they normally do to provide oxygen and remove carbon dioxide from the body. This can lead to a reduced amount of oxygen in the patient's bloodstream. Patients with ARDS are admitted to the intensive care unit (ICU) and need help with their breathing by being connected to a ventilator (breathing machine). ARDS can lead to injury in other organs of the body causing other problems but also death.

Over the past few years, reducing the size of each breath delivered by the ventilator in conjunction with the use of an occasional sustained deep breath called a "recruitment manoeuvre" have been used to try to prevent further damage to the lungs in people with ARDS. This ventilator strategy (termed the PHARLAP strategy) has been shown in a small research study to have some beneficial effects without causing any obvious harm, when compared to a current best practice ventilator strategy. The main beneficial effects of the PHARLAP strategy were to increase the amount of oxygen in the blood and to reduce markers of inflammation (the body reacting to a disease process) in the body. This study was too small to make a strong conclusion, so this study will be much larger and will assess whether patients who have developed ARDS are better off when we use the PHARLAP strategy. Three hundred and forty patients will be enrolled into this study in multiple ICUs across Australia and New Zealand.

The study hypothesis is that the PHARLAP strategy group will have a higher number of ventilator free days at day 28 than the control group.

DETAILED DESCRIPTION:
340 adult patients who have developed ARDS within the last 72 hours (and within 10 days of commencing mechanical ventilation) will be enrolled in 25- 30 intensive care units (ICUs) and randomly allocated to either the PHARLAP or a control ventilation strategy. PHARLAP strategy: Pressure control ventilation to maintain tidal volume 4-6 ml/kg and plateau pressure ≤ 30 cmH2O while tolerating respiratory acidosis if pH > 7.15; daily staircase recruitment manoeuvre and individualised Positive-end expiratory pressure (PEEP) titration.

Control strategy: Mechanical ventilation based on the ARDSnet protocol with tidal volume 6 ml/kg, plateau pressure ≤ 30 cmH2O and fraction inspired oxygen (FiO2)/PEEP titration according to a FiO2/PEEP/oxygen saturation combination chart. This has been modified for Australian and New Zealand practice to allow pressure control and pressure support ventilation. A standardised weaning from mechanical ventilation guideline will be used in both groups

ELIGIBILITY:
Inclusion Criteria:

Adult ICU patients who met all of the following criteria:

* Currently intubated and receiving mechanical ventilation
* Within 72 Hours of a diagnosis of ARDS (moderate and severe) based on the following Berlin definition:
* Within 1 week of a known clinical insult or new or worsening respiratory symptoms
* Bilateral opacities on chest x-ray (CXR) which are not fully explained by effusions, lobar/lung collapse or nodules
* Respiratory failure not fully explained by cardiac failure or fluid overload
* Arterial oxygen pressure (PaO2)/FiO2 < 200mmHg with PEEP ≥ 5cmH2O

Exclusion Criteria:

* > 72 hours since diagnosis of ARDS
* > 10 days of continuous mechanical ventilation
* Barotrauma (pneumothorax, pneumomediastinum, subcutaneous emphysema or any intercostal catheter for the treatment of air leak)
* Significant chest trauma i.e. multiple rib fractures
* Active bronchospasm or a history of significant chronic obstructive pulmonary disease or asthma
* Clinical suspicion for significant restrictive lung disease (history of pulmonary fibrosis or suggestive pulmonary function tests)
* Moderate or severe traumatic brain injury, the presence of an intracranial pressure monitor, or any medical condition associated with a clinical suspicion of raised intracranial pressure
* Unstable cardiovascular status defined as sustained heart rate < 40 or > 140 bpm, ventricular tachycardia, or SBP < 80mmHg
* Pregnancy
* Receiving ECMO
* Receiving high frequency oscillatory ventilation
* Death is deemed imminent and inevitable
* The treating physician believes it is not in the best interest of the patient to be enrolled in the trial
* Consent not obtained or refused by patient's legal surrogate

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2012-10; Primary Completion 2017-10 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Hodgson, PhD, FACP, BAppSc, Study Chair — Australian and New Zealand Intensive Care Research Centre (ANZIC-RC); Alistair Nichol, PhD, FCICM, Study Chair — Australian and New Zealand Intensive Care Research Centre (ANZIC-RC)
Locations (27):
- Australia (8):
  - Albury/Wodonga, Albury, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Royal Prince Alfred, Sydney, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - Flinders Medical Centre, Adelaide, South Australia
  - Geelong Hospital, Geelong, Victoria
  - The Alfred Hosptial, Melbourne, Victoria
- Ireland (5):
  - Adelaide and Meath (Tallaght) Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St Vincents Hospital, Dublin
  - University Hospital Limerick, Limerick
- New Zealand (3):
  - Middlemore Hospital, Otahuhu, Auckland
  - Auckland City Hospital (DCCM), Auckland
  - Auckland City Hospital CVICU, Auckland
- King Abdulaziz Medical City, Riyadh, Saudi Arabia
- United Kingdom (10):
  - Peterborough City Hospital, Peterborough, Cambridgeshire
  - Derriford Hospital, Plymouth, Devon
  - Princess Royal University Hospital, Orpington, Kent
  - Royal Surrey County Hospital, Guildford, Surrey
  - Southmead Hospital, Bristol
  - Hull Royal Infirmary, Hull
  - King's College Hospital, London
  - North Middlesex University Hospital, London
  - University Hospital, Lewisham, London
  - James Cook University Hospital, Middlesbrough

IPD SHARING:
Plan to Share IPD: Yes
The Australian and New Zealand Intensive Care Research Centre (ANZIC RC), Monash University supports the view that:
  * Publicly funded research data should be made available with as few restrictions as possible
  * Data sharing could enhance public well-being by maximising utilisation of gained knowledge, reducing redundant research and facilitating scientific innovation,
  * Data sharing must be responsible, recognise legal, regulatory, ethical and commercial constraints.
  The ANZIC-RC has formulated a policy and process to allow appropriate and responsible sharing of research data including prospective and completed studies.
  This Policy was guided by, Institute of Medicine principles for responsible sharing of clinical trial data:
  * Maximise the benefits of clinical trials
  * Minimising the risks of data sharing
  * Respect individual participants
  * Increase public trust in clinical trials
  * Conduct the sharing of trial data in a fair manner
  * Appropriately manage conflicts of interest.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Is available on request
Access Criteria: request made to custodian via Australian and New Zealand Intensive Care Research Centre
  See ANZIC-RC website term of reference document
URL: https://www.monash.edu/medicine/sphpm/anzicrc/governance

REFERENCES:
- [Background] Hodgson CL, Cooper DJ, Arabi Y, King V, Bersten A, Bihari S, Brickell K, Davies A, Fahey C, Fraser J, McGuinness S, Murray L, Parke R, Paul E, Tuxen D, Vallance S, Young M, Nichol A. Maximal Recruitment Open Lung Ventilation in Acute Respiratory Distress Syndrome (PHARLAP). A Phase II, Multicenter Randomized Controlled Clinical Trial. Am J Respir Crit Care Med. 2019 Dec 1;200(11):1363-1372. doi: 10.1164/rccm.201901-0109OC. PMID 31356105
- [Background] Hodgson C, Cooper DJ, Arabi Y, Bennett V, Bersten A, Brickell K, Davies A, Fahey C, Fraser J, McGuinness S, Murray L, Parke R, Tuxen D, Vallance S, Young M, Nichol AD; PHARLAP Study Investigators and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Permissive Hypercapnia, Alveolar Recruitment and Low Airway Pressure (PHARLAP): a protocol for a phase 2 trial in patients with acute respiratory distress syndrome. Crit Care Resusc. 2018 Jun;20(2):139-149. PMID 29852853
- [Background] Bihari S, Bersten A, Paul E, McGuinness S, Dixon D, Sinha P, Calfee CS, Nichol A, Hodgson C; PHARLAP Study Investigators. Acute respiratory distress syndrome phenotypes with distinct clinical outcomes in PHARLAP trial cohort. Crit Care Resusc. 2023 Oct 18;23(2):163-170. doi: 10.51893/2021.2.oa3. eCollection 2021 Jun. PMID 38045528

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PHARLAP Ventilation Group | Control Group Ventilation
Started | 58 | 57
Completed | 57 | 56
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- PHARLAP Intervention Arm: PHARLAP strategy (21) included pressure control mode, Tidal Volume (VT) of 4-6 ml/kg, and plateau airway pressures <28cm H2O (online supplement). Patients underwent daily maximal RMs with PEEP titration (a combined open lung procedure [COLP]) for up to the first 5 days The COLP was performed as follows. A staircase RM (SRM) was applied in pressure control ventilation at 15 6 3 cm H2O, with the PEEP increased to 20 cm H2O, then 30 cm H2O, and then 40 cm H2O for 2 minutes each. This step was followed by decremental PEEP titration from 25 cm H2O in 2.5-cm H2O steps for 3 minutes until the SpO2 decreased by 2% or more or to a minimum of 15 cm H2O PEEP if desaturation did not occur. Last, a brief RM returned the PEEP to a level 2.5 cm H2O above the level of desaturation. Airway pressures were minimized with permissive hypercapnia and targeting VT and plateau pressures ,6 ml/kg and ,28 cm H2O, respectively. Brief RMs could be performed throughout the day in case of hypoxemia (online supplement). The study's weaning protocol included daily assessments to identify patients who met weaning criteria and were suitable for a spontaneous breathing trial (online supplement) (24). After a successful spontaneous breathing trial, the ICU clinician reviewed the patient with a view to prompt extubation.
- Control Group: patients were ventilated according to the Acute Respiratory Distress Syndrome Network's low-VT/low PEEP ventilation protocol (4), including volume control mode, VT of 6 ml/kg, plateau airway pressures <30 cm H2O, and the low PEEP strategy (Table E2). RMs were not permitted.
- Total: Total of all reporting groups
Arm/Group | PHARLAP Intervention Arm | Control Group | Total
Number analyzed (Participants) | 58 | 56 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (14.0) | 53.2 (14.4) | 53.7 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 48
  Male | 36 | 30 | 66
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
APACHE II score [Median (Standard Deviation); unit: units on a scale] — Acute Physiology and Chronic Health Evaluation II (APACHE II) is a measure of disease severity derived from 3 scores: A) Physiology Score, 12 physiological variables assigned values between 0 (normal) and 4 (high or low abnormal range); B) Age; ranging 0 (44yrs or less) to 6 (75yrs or more); and C) Chronic Health; based on patients medical history with values from 0 (no history) to 5 (non-operative or emergency post-operative patients). Sub-scales are added to determine an overall score between 0 and 71, with increasing scores indicating increased risk of hospital death
  units on a scale | 23.2 (6.8) | 22.3 (7.7) | 22.8 (7.2)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.3 (10.1) | 30.3 (7.2) | 30.8 (8.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Ventilator Free Days at Day 28 Post Randomisation
Description: This is the total number of days calculated from day 1 (randomisation) to day 28 on which the patient was alive and received no assistance from invasive mechanical ventilation. Scores range between 0 (no ventilator free days) to 28 (no days on ventilator).
Time Frame: 28 days post randomisation
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | PHARLAP Ventilation Group | Control Group Ventilation
Number analyzed (Participants) | 57 | 56
days | 16 [0 to 21] | 14.5 [0 to 21.5]

2. Secondary Outcome: PaO2/FiO2 Ratio and Static Lung Compliance
Description: PaO2/FiO2 ratio is the ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen (FiO2 expressed as a fraction, not a percentage). ARDS severity Mild 200-300 / Moderate 100-200 / Severe <100.
Time Frame: Up to day 28 post randomisation
Reporting Status: Not Posted, anticipated posting 2025-01

3. Secondary Outcome: Baseline to Day 3 Change in IL-8 and IL-6 Concentrations in Broncho-alveolar Lavage and Plasma
Description: IL-8 is an important protein related to inflammation, Interleukin (IL)-6 is produced at the site of inflammation and plays a key role in the acute phase response
Time Frame: Day 3 post randomisation
Reporting Status: Not Posted, anticipated posting 2025-01

4. Secondary Outcome: Number of Severe Hypotension Events
Description: Hypotension requiring increased vasopressor Days 1-28
Time Frame: Up to 28 days post randomisation
Measure: Number; unit: events
Arm/Group | PHARLAP Ventilation Group | Control Group Ventilation
Number analyzed (Participants) | 57 | 56
events | 20 | 12

5. Secondary Outcome: Number of Participants With Barotrauma
Description: Evidence of Pneumothorax requiring Drainage
Time Frame: Up to 90 days post randomisation
Measure: Count of Participants; unit: Participants
Arm/Group | PHARLAP Ventilation Group | Control Group Ventilation
Number analyzed (Participants) | 57 | 56
Participants | 3 | 2

6. Secondary Outcome: Use of Rescue Therapies for Severe Hypoxaemia - Inhaled Nitric Oxide, Inhaled Prostacyclin, Prone Positioning, High Frequency Oscillatory Ventilation and Extracorporeal Membrane Oxygenation (ECMO)
Description: The use of various rescue therapies (each of the therapies is compared between groups - per patient). the various therapies measured are inhaled nitric oxide, inhaled prostacyclin, prone positioning, high frequency oscillatory ventilation and extracorporeal membrane oxygenation (ECMO)
Time Frame: Within hospital admission
Reporting Status: Not Posted, anticipated posting 2025-01

7. Secondary Outcome: Mortality
Description: At timepoints: day 28
Time Frame: at day 28
Measure: Count of Participants; unit: Participants
Arm/Group | PHARLAP Ventilation Group | Control Group Ventilation
Number analyzed (Participants) | 57 | 56
Participants | 14 | 15

8. Secondary Outcome: ICU Length of Stay
Description: The number of days a person stayed in the ICU. A fraction of a day is considered a day
Time Frame: From admission to ICU up to 6 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | PHARLAP Ventilation Group | Control Group Ventilation
Number analyzed (Participants) | 57 | 56
days | 11.1 [6.2 to 20.1] | 13.8 [6.8 to 22.5]

9. Secondary Outcome: Incidence of Acute Kidney Injury (AKI)
Description: The incidence of Acute Renal Injury - measured by the use of Continuous Renal Replacement Therapy (CRRT) in each person
Time Frame: Within hospital admission
Reporting Status: Not Posted, anticipated posting 2025-01

10. Secondary Outcome: Quality of Life Assessment
Description: SF36v2 will be used Medical Outcomes Study. Scoring the RAND is a two-step process. First, pre-coded numeric values are recoded. Note that all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores.
Time Frame: 6 months post randomisation
Reporting Status: Not Posted, anticipated posting 2025-01

11. Secondary Outcome: Cost Effectiveness Analysis
Description: This will be based on EQ-5D. EQ-5D is the most widely used health-related quality of life questionnaire in health economic evaluations.[62] EQ-5D can be used to derive a set of values that reflect people's opinions of the relative importance of different health problems. These values can be used to derive QALYs for application in cost-effectiveness and cost-utility evaluations.
Time Frame: 6 months post randomisation
Reporting Status: Not Posted, anticipated posting 2025-01

12. Secondary Outcome: Hospital Length of Stay
Description: The length of time in days a participant stayed in hospital. A fraction of a day is considered 1 day.
Time Frame: From admission up to 6 months
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | PHARLAP Ventilation Group | Control Group Ventilation
Number analyzed (Participants) | 57 | 56
Days | 20.1 [8.1 to 37.2] | 17.9 [9.0 to 39.0]

ADVERSE EVENTS:
Time Frame: Adverse events will be collected from randomisation up until the 90 day follow up, up to 90 days in total
Description: Patients with critical illness and ARDS will experience a number of common aberrations in lab values, signs and symptoms due to the severity of underlying illness and the impact of standard therapies. These do not necessarily constitute an adverse event unless they require significant intervention or are of concern in the investigator's clinical judgement.
  Primary outcome data (all-cause mortality) not available for one participant in the intervention group, drew to withdrawn consent
Arm/Group | PHARLAP Ventilation Group | Control Group Ventilation
All-Cause Mortality (participants affected / at risk) | 14/57 | 17/56
Serious Adverse Events (participants affected / at risk) | 23/58 | 15/56
Other Adverse Events (participants affected / at risk) | 9/58 | 4/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PHARLAP Ventilation Group (N=58) | Control Group Ventilation (N=56)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 3 — Requiring chest tube
Severe Hypotension (Cardiac disorders) | 20 | 12 — requiring a change in vasopressors
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PHARLAP Ventilation Group (N=58) | Control Group Ventilation (N=56)
refractory acidosis (Metabolism and nutrition disorders) | 9 | 4 — acidosis refractory to normal mangament

LIMITATIONS AND CAVEATS:
The power of the study was limited by lower than expected recruitment rates, early termination of the trial (due to the publication of the ART trial), and treatment crossovers. Blinding was not possible within the ICU, staff and relatives were aware of group allocation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-11-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT01667146/Prot_SAP_000.pdf
  • Informed Consent Form (2013-09-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT01667146/ICF_001.pdf